CLINICAL TRIAL: NCT00215579
Title: Determining the Effects of Risperdal Consta in Patients With Psychotic Disorders and Incomplete Adherence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5631; RIS-SCH-421 (Other: Study specific ID)
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2012-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Depot Risperidone Microsphere (Consta)

SUMMARY:
As many as 75 percent of patients with schizophrenia have difficulty taking their oral medication on a regular basis. This may lead to worsening of symptoms. Clinicians commonly respond to these problems by adding adjunctive medications, despite the absence of systematic studies that support such practices. It is possible, however, that in many of these cases, the unstable course and/or unsatisfactory treatment response reflects incomplete adherence with the originally prescribed oral antipsychotic, rather than a need for adjunctive medications. This study will examine whether switching patients who demonstrate an unstable course and/or an unsatisfactory clinical response to a long-acting injectable preparation as the primary antipsychotic may enhance medication adherence and improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be male or female
* Between 18-65 years of age and will meet DSM-IV criteria for schizophrenia or schizoaffective disorder.
* The subject must have, in their physicians opinion, an unstable course and must have been treated with an oral antipsychotic.

Exclusion Criteria:

* Pregnant and breast feeding females will be excluded.
* Because fluoxetine is known to change the plasma level of CONSTA, subjects taking fluoxetine within two weeks of starting the study will be excluded.
* Patients who are known to have a hypersensitivity to oral Risperdal will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2004-04; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William H Wilson, PhD, Principal Investigator — Duke University
Locations (1):
- John Umstead Hospital, Butner, North Carolina, United States